CLINICAL TRIAL: NCT03457610
Title: Speech Therapy in the Management of Difficult-to-treat Chronic Cough
Brief Title: Speech Therapy in the Management of Chronic Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marta Dąbrowska, Principal Investigator, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pulm2017
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Cough; Speech Therapy
Keywords: chronic cough; speech and language intervention; difficult-to-treat cough
MeSH Terms: conditions — Cough; Communication Disorders; Chronic Cough; Speech | interventions — Speech Therapy

STUDY DESIGN:
Intervention Model Description: prospective, single arm, single center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Speech and language intervention (Experimental)
  Interventions: Behavioral: Speech and language intervention

INTERVENTIONS:
Behavioral: Speech and language intervention — Speech therapy includes education about cough and vocal hygiene, teaching strategies to reduce cough, breathing and vocal exercises. The whole therapy consists of eight sessions once a week.
  Other Names: Speech therapy; Voice therapy

SUMMARY:
Speech and language intervention (speech therapy) is one of the few methods which seem to be useful in management of persistent chronic cough. This method has not been available for patients with cough in Poland so far.The aim of the study is to implement speech therapy to the management plan of patients with difficult-to-treat chronic cough and to analyze its efficacy in this particular group.

Patients with difficult-to treat chronic cough will be offered speech and language intervention as an added therapy. The effectiveness of speech therapy will be measured by changes in cough severity, its influence on quality of life and cough challenge test before and after speech therapy measured in every patient.

DETAILED DESCRIPTION:
The efficacy of management of chronic cough in adults is limited. Speech and language intervention (speech therapy) is one of the few methods which seem to be useful in management of persistent chronic cough. This method has not been available for patients with cough in Poland so far.

The aim of the study is to implement speech therapy to the management plan of patients with difficult-to-treat chronic cough and to analyze its efficacy in this particular group.

Patients, who are diagnosed and unsuccessfully managed because of difficult-to treat chronic cough, will be offered speech and language intervention as an added therapy. It is based on the technique described by Vertigan et al.The entire therapy will consist of eight sessions once a week.

Cough severity, its influence on quality of life and cough challenge test with capsaicin will be assessed by Visual Analogue Scale, Leicester Cough Questionnaire and cough challenge test with capsaicin will be performed before and after speech therapy in every patient to analyze its effectiveness

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 80 years,
2. chronic cough lasting more than six months
3. earlier thorough diagnosing of cough reason
4. unsuccessful cough management despite at least 3 months of earlier treatment
5. no symptoms of any airway infection during last 4 weeks.

Exclusion Criteria:

1. lack of opportunity to participate in speech therapy sessions
2. cough lasting less than 6 months
3. active cigarette smoking
4. taking ACE inhibitors
5. symptoms of airway infection (other than cough).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Cough severity | 3 months
  measured by Visual Analogue Scale (VAS), range 0-100 mm, the more severe cough , the higher value in VAS score

SECONDARY OUTCOMES:
Cough related quality of life | 3 months
  measured by Leicester Cough Questionnaire (LCQ)- health related Quality of Life Questionnaire dedicaated for patients, who cough; rangeof total LCQ is 3 to 21 points; higher values represent less intense cough
Sensitivity of cough reflex | 3 months
  measured by cough challenge test with capsaicin

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Pneumonology and Allergology, Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Background] Morice AH, Fontana GA, Belvisi MG, Birring SS, Chung KF, Dicpinigaitis PV, Kastelik JA, McGarvey LP, Smith JA, Tatar M, Widdicombe J; European Respiratory Society (ERS). ERS guidelines on the assessment of cough. Eur Respir J. 2007 Jun;29(6):1256-76. doi: 10.1183/09031936.00101006. No abstract available. PMID 17540788
- [Background] Vertigan AE, Theodoros DG, Gibson PG, Winkworth AL. Efficacy of speech pathology management for chronic cough: a randomised placebo controlled trial of treatment efficacy. Thorax. 2006 Dec;61(12):1065-9. doi: 10.1136/thx.2006.064337. Epub 2006 Jul 14. PMID 16844725
- [Result] Gibson P, Wang G, McGarvey L, Vertigan AE, Altman KW, Birring SS; CHEST Expert Cough Panel. Treatment of Unexplained Chronic Cough: CHEST Guideline and Expert Panel Report. Chest. 2016 Jan;149(1):27-44. doi: 10.1378/chest.15-1496. Epub 2016 Jan 6. PMID 26426314